CLINICAL TRIAL: NCT03712787
Title: An Extension Study of ABBV-8E12 in Early Alzheimer's Disease
Brief Title: An Extension Study of ABBV-8E12 in Early Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Discontinued because of lack of efficacy in the parent study (Study M15-566; NCT02880956).
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-570; 2018-000268-26 (EudraCT Number)
Record Dates: First submitted 2018-10-18; First posted 2018-10-19 (Actual); Results first posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-08

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tilavonemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 300 mg/1000 mg Tilavonemab (Experimental): Participants who received 300 mg tilavonemab in Study M15-566 receive 1000 mg tilavonemab in Study M15-570 via intravenous (IV) infusion every 4 weeks for up to 5.5 years.
  Interventions: Drug: Tilavonemab
- 1000 mg/1000 mg Tilavonemab (Experimental): Participants who received 1000 mg tilavonemab in Study M15-566 continue on the same dose in Study M15-570 via IV infusion every 4 weeks for up to 5.5 years.
  Interventions: Drug: Tilavonemab
- 2000 mg/2000 mg Tilavonemab (Experimental): Participants who received 2000 mg tilavonemab in Study M15-566 continue on the same dose in Study M15-570 via IV infusion every 4 weeks for up to 5.5 years.
  Interventions: Drug: Tilavonemab
- PBO/2000 mg Tilavonemab (Experimental): Participants who received placebo (PBO) in Study M15-566 receive 2000 mg tilavonemab in Study M15-570 via IV infusion every 4 weeks for up to 5.5 years.
  Interventions: Drug: Tilavonemab

INTERVENTIONS:
Drug: Tilavonemab — solution for IV infusion
  Other Names: ABBV-8E12

SUMMARY:
The purpose of this study is to assess the long-term safety and tolerability of ABBV-8E12 in participants with early AD.

ELIGIBILITY:
Inclusion Criteria:

* All subjects with early AD who complete Study M15-566 (NCT02880956), meet all inclusion criteria, and do not meet any exclusion criteria are eligible for enrollment
* Subject was compliant during participation in Study M15-566 (NCT02880956)
* Subject has an identified, reliable study partner who has frequent contact with the subject and who will provide information as to the subject's cognitive and functional abilities

Exclusion Criteria:

* The subject has any significant change in his/her medical condition since participation in Study M15-566 (NCT02880956) that could interfere with the subject's participation in Study M15-570, could place the subject at increased risk, or could confound interpretation of study results
* More than 8 weeks have elapsed since the subject received his/her last dose of study drug in Study M15-566 (NCT02880956)
* The subject is concurrently enrolled in another interventional clinical study involving a therapeutic agent with the exception of Study M15-566 (NCT02880956)

Ages: 57 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Actual)
Dates: Start 2019-03-22 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (57):
- United States (32):
  - Banner University of Arizona Medical Center Phoenix /ID# 203959, Phoenix, Arizona
  - Irvine Clinical Research /ID# 204000, Irvine, California
  - Ucsd /Id# 204001, La Jolla, California
  - University of California, San /ID# 204011, San Francisco, California
  - Brain Matters Research /ID# 203957, Delray Beach, Florida
  - Neuropsychiatric Research Center of Southwest Florida /ID# 203956, Fort Myers, Florida
  - Mayo Clinic /ID# 203995, Jacksonville, Florida
  - Synexus Clinical Research US, Inc. /ID# 203992, Orlando, Florida
  - University of South Florida /ID# 204009, Tampa, Florida
  - Synexus Clinical Research US, Inc /ID# 204010, The Villages, Florida
  - Emory University / Emory Brain Health Center /ID# 203999, Atlanta, Georgia
  - NeuroStudies.net, LLC /ID# 204004, Decatur, Georgia
  - Advocate Lutheran General Hospital /ID# 203993, Park Ridge, Illinois
  - Southern IL Univ School of Med /ID# 203952, Springfield, Illinois
  - Indiana University /ID# 203989, Indianapolis, Indiana
  - University of Kansas Medical Center - Alzheimer's Disease Center /ID# 203960, Fairway, Kansas
  - University of Kentucky Chandler Medical Center /ID# 203996, Lexington, Kentucky
  - Massachusetts General Hospital /ID# 203954, Boston, Massachusetts
  - Brigham and Women's Physicians /ID# 204003, Boston, Massachusetts
  - Hattiesburg Clinic /ID# 213435, Hattiesburg, Mississippi
  - Princeton Medical Institute /ID# 203953, Princeton, New Jersey
  - North Shore University Hospital /ID# 203994, New Hyde Park, New York
  - Duke Univ Med Ctr /ID# 203958, Durham, North Carolina
  - Oregon Health and Science University /ID# 203997, Portland, Oregon
  - Keystone Clinical Studies LLC /ID# 213183, Plymouth Meeting, Pennsylvania
  - Rhode Island Hospital /ID# 204005, Providence, Rhode Island
  - Vanderbilt Ingram Cancer Center /ID# 203951, Nashville, Tennessee
  - Kerwin Research Center /ID# 203998, Dallas, Texas
  - Houston Methodist Hospital /ID# 204002, Houston, Texas
  - McGovern Medical School /ID# 213312, Houston, Texas
  - University of Utah /ID# 203991, Salt Lake City, Utah
  - Integrated Neurology Services /ID# 203990, Alexandria, Virginia
- Australia (4):
  - St Vincent's Centre for Applied Medical Research /ID# 204903, Darlinghurst, New South Wales
  - Griffith University /ID# 204905, Southport, Queensland
  - Austin Health /ID# 204906, Heidelberg, Victoria
  - Australian Alzheimer's Res Fou /ID# 204904, Nedlands, Western Australia
- Belgium (3):
  - UCL Saint-Luc /ID# 204963, Woluwe-Saint-Lambert, Brussels Capital
  - Universitair Ziekenhuis Leuven /ID# 204965, Leuven, Vlaams-Brabant
  - Groupe Sante CHC - Clinique du MontLegia /ID# 204964, Liège
- Canada (2):
  - Parkwood Institute /ID# 204121, London, Ontario
  - Toronto Memory Program /ID# 204120, Toronto, Ontario
- Rigshospitalet /ID# 204591, Copenhagen Ø, Capital Region, Denmark
- Finland (2):
  - Clinical Research Services Turku /ID# 205924, Turku, Southwest Finland
  - Ita-Suomen Yliopisto /ID# 204538, Kuopio
- Italy (6):
  - AOU di Modena /ID# 203904, Modena, Emilia-Romagna
  - Policlinico Agostino Gemelli /ID# 203906, Rome, Lazio
  - Azienda Ospedaliera di Perugia /ID# 203905, Perugia, Umbria
  - IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli /ID# 203903, Brescia
  - Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 203902, Milan
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 203901, Milan
- CGM Research Trust /ID# 204907, Burwood, New Zealand
- Spain (4):
  - Fundacion CITA Alzheimer Fundazioa /ID# 204521, Donostia / San Sebastian, Basque Country
  - Fundacio ACE /ID# 204520, Barcelona
  - Hospital Clinic de Barcelona /ID# 204519, Barcelona
  - Hospital Universitario 12 de Octubre /ID# 204518, Madrid
- Sweden (2):
  - Karolinska University Hospital Huddinge /ID# 203900, Stockholm, Stockholm County
  - Sahlgrenska University Hospital Molndal /ID# 203899, Mölndal, Västra Götaland County

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 364 participants who had completed the parent study (Study M15-566; NCT02880956) were enrolled into this extension study from a total of 57 sites in the United States, Australia, Belgium, Canada, Denmark, Finland, Italy, New Zealand, Spain, and Sweden.
Pre-assignment Details: Prior to enrollment, 87 participants had received tilavonemab 300 mg, 97 participants had received tilavonemab 1000 mg, 88 participants had received tilavonemab 2000 mg, and 92 participants had received placebo in the parent study.
  One enrolled participant did not receive any study drug and was not included in any analysis.
Groups:
- 300 mg/1000 mg Tilavonemab: Participants who received 300 mg tilavonemab in Study M15-566 received 1000 mg tilavonemab in Study M15-570 via intravenous (IV) infusion every 4 weeks.
- 1000 mg/1000 mg Tilavonemab: Participants who received 1000 mg tilavonemab in Study M15-566 were continued on the same dose in Study M15-570 via IV infusion every 4 weeks.
- 2000 mg/2000 mg Tilavonemab: Participants who received 2000 mg tilavonemab in Study M15-566 were continued on the same dose in Study M15-570 via IV infusion every 4 weeks.
- PBO/2000 mg Tilavonemab: Participants who received placebo (PBO) in Study M15-566 received 2000 mg tilavonemab in Study M15-570 via IV infusion every 4 weeks.
Period: Overall Study
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab
Started (enrolled and treated) | 87 | 97 | 88 | 91
Completed | 0 | 0 | 0 | 0
Not Completed | 87 | 97 | 88 | 91
Not completed — Adverse Event | 2 | 3 | 0 | 4
Not completed — Withdrawal by Subject | 4 | 14 | 12 | 8
Not completed — Lost to Follow-up | 1 | 1 | 2 | 1
Not completed — COVID-19 Logistical Restrictions | 1 | 1 | 0 | 0
Not completed — COVID-19 Infection | 0 | 1 | 0 | 0
Not completed — Other, Not Specified | 79 | 77 | 74 | 78

BASELINE CHARACTERISTICS:
Population: Safety Data Set: All participants who received at least 1 dose of study drug in M15-570.
Groups:
- 300 mg/1000 mg Tilavonemab: Participants who received 300 mg tilavonemab in Study M15-566 received 1000 mg tilavonemab in Study M15-570 via IV infusion every 4 weeks.
- PBO/2000 mg Tilavonemab: Participants who received PBO in Study M15-566 received 2000 mg tilavonemab in Study M15-570 via IV infusion every 4 weeks.
- Total: Total of all reporting groups
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab | Total
Number analyzed (Participants) | 87 | 97 | 88 | 91 | 363
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 8 | 11 | 14 | 10 | 43
  >= 65 years | 79 | 86 | 74 | 81 | 320
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 48 | 48 | 56 | 191
  Male | 48 | 49 | 40 | 35 | 172
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 1 | 0 | 2 | 6
  White | 81 | 94 | 86 | 89 | 350
  More than one race | 0 | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 3 | 4 | 16
  None | 82 | 93 | 85 | 87 | 347

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Discontinuation of Study Drug, and Fatal TEAEs
Description: Treatment emergent adverse events (TEAEs) are defined as any adverse event (AE) from the time of study drug administration until 20 weeks after discontinuation of study drug. An AE is defined as any untoward medical occurrence, which does not necessarily have a causal relationship with treatment. A serious AE (SAE) is defined as any event that: results in death; is life-threatening; results in hospitalization or prolongation of hospitalization; is a congenital anomaly; results in persistent or significant disability/incapacity; is an important medical event requiring medical or surgical intervention to prevent serious outcome. Severity of AEs was categorized as mild, moderate, or severe. Relationship of the AE to the study treatment was categorized as having a reasonable possibility or no reasonable possibility.
Time Frame: From first dose of study drug to 20 weeks after last dose of study drug; overall median time on treatment was 279 days.
Population: Safety Data Set: All participants who received at least 1 dose of study drug in Study M15-570.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab
Number analyzed (Participants) | 87 | 97 | 88 | 91
Participants
  Any TEAE | 54 | 66 | 59 | 57
  Severe TEAE | 9 | 8 | 10 | 7
  TEAE With a Reasonable Possibility of Relationship to Study Drug | 7 | 10 | 15 | 5
  Serious TEAE | 16 | 11 | 12 | 10
  TEAE Leading to Discontinuation of Study Drug | 2 | 4 | 0 | 5
  Fatal TEAE | 1 | 1 | 1 | 0

2. Primary Outcome: Hematology: Number of Participants With Postbaseline Potentially Clinically Significant (PCS) Values
Description: Clinical laboratory PCS criteria were adapted from National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Baseline to 20 weeks after last dose of study drug; overall median time on treatment was 279 days.
Population: Safety Data Set: All participants who received at least 1 dose of study drug in Study M15-570.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab
Number analyzed (Participants) | 87 | 97 | 88 | 91
Participants
  Hemoglobin - Low (< 100 g/L) | 1 | 0 | 2 | 1
  Hemoglobin - High (> 40 g/L above Upper Limit of Normal [ULN]) | 0 | 0 | 0 | 0
  Platelets - Low (< 75 × 10^9/L) | 0 | 0 | 0 | 0
  Leukocytes - Low (< 2 × 10^9/L) | 0 | 0 | 0 | 0
  Leukocytes - High (> 100 × 10^9/L) | 0 | 0 | 0 | 0
  Neutrophils - Low (< 1 × 10^9/L) | 1 | 0 | 0 | 0
  Lymphocytes - Low (< 0.5 × 10^9/L) | 0 | 0 | 1 | 0
  Lymphocytes - High (> 20 × 10^9/L) | 0 | 0 | 0 | 0
  Activated Partial Thromboplastin Time (> ULN) | 0 | 0 | 0 | 0
  Prothrombin International Normalized Ratio (> ULN) | 0 | 0 | 0 | 0

3. Primary Outcome: Clinical Chemistry: Percentage of Participants With Postbaseline PCS Values
Description: Clinical laboratory PCS criteria were adapted from NCI CTCAE version 4.03
Time Frame: Baseline to 20 weeks after last dose of study drug; overall median time on treatment was 279 days.
Population: Safety Data Set: All participants who received at least 1 dose of study drug in Study M15-570.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab
Number analyzed (Participants) | 87 | 97 | 88 | 91
Participants
  Alanine Aminotransferase (> 3 × ULN) | 0 | 0 | 0 | 0
  Aspartate Aminotransferase (> 3 × ULN) | 0 | 0 | 0 | 0
  Alkaline Phosphatase (> 2.5 × ULN) | 0 | 0 | 0 | 0
  Bilirubin (> 1.5 × ULN) | 0 | 0 | 1 | 1
  Creatinine (> 1.5 × ULN) | 0 | 0 | 0 | 0
  Calcium - Low (< 1.75 mmol/L) | 0 | 0 | 0 | 0
  Calcium - High (> 3.1 mmol/L) | 0 | 0 | 0 | 0
  Sodium - Low (< 130 mmol/L) | 0 | 1 | 0 | 1
  Sodium - High (> 155 mmol/L) | 0 | 0 | 0 | 0
  Potassium - Low (< 3 mmol/L) | 0 | 0 | 0 | 0
  Potassium - High (> 6 mmol/L) | 0 | 0 | 0 | 0
  Glucose - Low (< 2.2 mmol/L) | 0 | 0 | 0 | 0
  Glucose - High (> 13.9 mmol/L) | 0 | 0 | 0 | 1
  Albumin (< 20 g/L) | 0 | 0 | 0 | 0
  Cholesterol (> 12.92 mmol/L) | 0 | 0 | 0 | 0
  Triglycerides (> 5.7 mmol/L) | 0 | 0 | 1 | 0
  Phosphate (< 0.6 mmol/L) | 0 | 0 | 0 | 0
  Uric acid (> 590 μmol/L) | 0 | 0 | 0 | 0

4. Primary Outcome: Columbia-Suicide Severity Rating Scale (C-SSRS) During Double-Blind Treatment Period
Description: The C-SSRS is a systematically administered instrument developed to track suicidal adverse events across a treatment study. The instrument is designed to assess suicidal behavior and ideation, track and assess all suicidal events, as well as the lethality of attempts. Suicidal ideation categories include the following: wish to be dead; nonspecific active suicidal thoughts; active suicidal ideation without intent to act; active suicidal ideation with some intent to act but no plan; active suicidal ideation with plan and intent. Suicidal behavior categories include the following: actual attempt; interrupted attempt; aborted attempt; preparatory acts or behavior; suicidal behavior; completed suicide.
Time Frame: Baseline to 20 weeks after last dose of study drug; overall median time on treatment was 279 days.
Population: Safety Data Set: All participants who received at least 1 dose of study drug in Study M15-570.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab
Number analyzed (Participants) | 87 | 97 | 88 | 91
Participants
  Suicidal behaviors or ideations | 4 | 3 | 8 | 4
  Suicidal behaviors | 0 | 0 | 0 | 0
  Suicidal ideations | 4 | 3 | 8 | 4
  Suicidal ideations only (No Suicidal Behavior) | 4 | 3 | 8 | 4

5. Primary Outcome: Brain Magnetic Resonance Imaging (MRI) Results: Number of Participants With Cerebral Edemas, New Microhemorrhage(s), and Severe White Matter Disease
Time Frame: Baseline to 20 weeks after last dose of study drug; overall median time on treatment was 279 days.
Population: Safety Data Set: All participants who received at least 1 dose of study drug in Study M15-570. Participants with postbaseline value for the respective parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab
Number analyzed (Participants) | 79 | 84 | 79 | 78
Participants
  Cerebral Edemas | 1 | 1 | 0 | 0
  Questionable Cerebral Edemas | 0 | 1 | 0 | 0
  New Microhemorrhage(s) | 4 | 5 | 11 | 5
  Severe White Matter Disease | 9 | 5 | 6 | 5

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: an overall median of 353.5 days. Serious and Other Adverse Events: From first dose of study drug to 20 weeks after last dose of study drug; overall median time on treatment was 279 days.
Arm/Group | 300 mg/1000 mg Tilavonemab | 1000 mg/1000 mg Tilavonemab | 2000 mg/2000 mg Tilavonemab | PBO/2000 mg Tilavonemab
All-Cause Mortality (participants affected / at risk) | 2/87 | 1/97 | 1/88 | 0/91
Serious Adverse Events (participants affected / at risk) | 16/87 | 11/97 | 12/88 | 10/91
Other Adverse Events (participants affected / at risk) | 26/87 | 37/97 | 33/88 | 26/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg/1000 mg Tilavonemab (N=87) | 1000 mg/1000 mg Tilavonemab (N=97) | 2000 mg/2000 mg Tilavonemab (N=88) | PBO/2000 mg Tilavonemab (N=91)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CARDIOPULMONARY FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETINAL ARTERY OCCLUSION (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BILIARY COLIC (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
CYSTITIS ESCHERICHIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONIA LEGIONELLA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL INTESTINAL PERFORATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SOFT TISSUE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLORECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DEMENTIA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BEHAVIOUR DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
AORTIC STENOSIS (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 300 mg/1000 mg Tilavonemab (N=87) | 1000 mg/1000 mg Tilavonemab (N=97) | 2000 mg/2000 mg Tilavonemab (N=88) | PBO/2000 mg Tilavonemab (N=91)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 5 (6) | 3 (3) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 4 (10) | 8 (8) | 0 (0) | 1 (3)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 6 (8) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 10 (14) | 10 (12) | 12 (16) | 10 (13)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 6 (6) | 2 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (6) | 4 (4) | 3 (3) | 5 (7)
DIZZINESS (Nervous system disorders) | 5 (5) | 2 (2) | 2 (2) | 2 (3)
AGITATION (Psychiatric disorders) | 1 (1) | 6 (6) | 2 (3) | 0 (0)
ANXIETY (Psychiatric disorders) | 3 (3) | 1 (1) | 7 (8) | 3 (3)
CONFUSIONAL STATE (Psychiatric disorders) | 1 (1) | 2 (2) | 4 (4) | 5 (6)
DELUSION (Psychiatric disorders) | 0 (0) | 1 (1) | 5 (5) | 2 (2)
HYPERTENSION (Vascular disorders) | 2 (2) | 5 (5) | 5 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
Study M15-570 was discontinued because of lack of efficacy in the parent study (Study M15-566) and 2) the tilavonemab development program was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03712787/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-30): https://cdn.clinicaltrials.gov/large-docs/87/NCT03712787/SAP_001.pdf